#### **Study Document Cover Page**

Official Title: Brain Dynamic Audio Stimulation for Improving Sleep Quality and Circadian

Rhythm in Healthcare Workers

**Short Title:** Brain Dynamic Audio Stimulation

**Document Type:** Statistical Analysis Plan **IRB Number:** CMMC IRB No. 11404-012

Organization Name: Chi Mei Medical Center (CMMC)

Principal Investigator: Hong-Min, Lin

**Document Date: 2026-01-01** 

Version: 2.0

Confidentiality Statement: This document contains confidential information intended for

regulatory and research purposes only.

#### Statistical Analysis Plan (SAP)

Study Title: Effectiveness of Brain Dynamic Audio Stimulation for Improving Insomnia

and Sleep Cycles in Healthcare Professionals (BDAS-HP)

**Protocol No.:** 11404-012

Version: 2.0

Date: January 1, 2026

**Sponsor/Institution:** Chi-Mei Medical Center **Principal Investigator:** Dr. Hong-Min Lin

## 1. Analysis Objectives and Endpoints

### 1.1 Primary Objective

To evaluate the effect of Brain Dynamic Audio Stimulation (BDAS) on insomnia severity as measured by the **Insomnia Severity Index (ISI)** before and after a two-week intervention.

### 1.2 Secondary Objectives

To assess the effect of BDAS on objective sleep-related parameters, including:

- Sleep onset success rate
- Sleep onset latency
- Sleep efficiency
- Short-term sleep stage distribution derived from EEG-based hypnograms

#### 1.3 Endpoints

#### **Primary Endpoint**

 Mean change in total ISI score from baseline (pre-intervention) to post-intervention (after 2 weeks)

#### **Secondary Endpoints**

- Sleep onset success rate following BDAS exposure
- Mean sleep onset latency (seconds) before and after 2 weeks of BDAS use
- Mean sleep efficiency (%) before and after BDAS intervention
- Proportion of time spent in each sleep stage (Wake, N1, N2, N3, REM) during EEG recording sessions

## 2. Analysis Populations

| Population | Definition |
|---|---|
| Full Analysis Set | All participants who received at least one BDAS session |
| (FAS) | and provided baseline ISI data |
| Per-Protocol Set | Participants completing ≥80% of BDAS sessions without major |
| (PPS) | protocol deviations |
| Safety Set | All participants who initiated BDAS intervention |

- Primary analyses will be conducted on the FAS
- Sensitivity analyses will be performed using the **PPS**

## 3. General Statistical Principles

- All statistical analyses will be conducted using SPSS (v28 or later) or R (v4.3 or later)
- All tests will be **two-tailed**
- Statistical significance will be defined as p < 0.05
- Continuous variables will be summarized as:
  - $\circ$  Mean  $\pm$  standard deviation (SD), or
  - o Median and interquartile range (IQR) if non-normally distributed
- Categorical variables will be summarized as counts and percentages
- Normality will be assessed using Shapiro-Wilk tests and visual inspection (Q-Q plots)

# 4. Handling of Missing Data

- For ISI analysis, participants with both baseline and post-intervention data will be included
- No imputation will be performed for missing objective sleep measures
- Sensitivity analyses excluding incomplete cases will be conducted to assess robustness

version:2

### 5. Statistical Methods

#### 5.1 Primary Analysis: ISI Score

- Paired-sample t-test will be used to compare pre- and post-intervention ISI scores
- If normality assumptions are violated, the Wilcoxon signed-rank test will be applied
- Effect sizes will be reported using:
  - o Cohen's d
  - o Hedges' g
- Mean difference with 95% confidence intervals (CI) will be presented

### 5.2 Secondary Analysis: Sleep Onset Success Rate

- Sleep onset success will be defined as transition from wakefulness to any sleep stage during the recording period
- Success rates will be summarized descriptively as proportions (%)
- No inferential testing is planned due to the exploratory nature of this endpoint

### 5.3 Secondary Analysis: Sleep Onset Latency

- Sleep onset latency is defined as time (seconds) from recording start to first epoch of sleep
- **Independent-sample t-tests** will be used to compare latency between:
  - o Initial use
  - o After 2 weeks of BDAS use
- Each sleep session will be treated as an independent observation to maximize statistical power
- Effect sizes will be reported using Cohen's d and Hedges' g

#### 5.4 Secondary Analysis: Sleep Efficiency

- Sleep efficiency is defined as: (Total sleep time / total recording time) × 100%
- Independent-sample t-tests will be used to compare sleep efficiency before and after BDAS intervention
- Effect sizes (Cohen's d, Hedges' g) and 95% CIs will be reported

### 5.5 Exploratory Analysis: Sleep Stage Distribution

- Sleep stages will be classified according to AASM criteria
- Proportion of time spent in each stage (Wake, N1, N2, N3, REM) will be summarized descriptively
- Where appropriate, paired-sample t-tests or Wilcoxon tests will be applied for exploratory comparisons
- Results will be interpreted descriptively due to short recording duration

## 6. Outlier and Data Quality Management

- Outliers (>3 SD from the mean) will be reviewed against raw EEG and recording logs
- Artifactual recordings (movement, muscle noise) will be excluded prior to analysis
- A minimum of 80% usable recording time is required for inclusion in EEG-based analyses

## 7. Sample Size Considerations

- This study is exploratory in nature
- Based on prior observations of ISI improvement (mean reduction ≈5 points, SD ≈4), a sample size of 15 participants provides sufficient power to detect large within-subject effects
- No formal hypothesis-driven power calculation is applied for secondary outcomes

### 8. Interim and Sensitivity Analyses

- No interim analyses are planned
- Sensitivity analyses will include:
  - Reanalysis excluding identified outliers
  - o Non-parametric alternatives where appropriate
  - PPS-based comparisons

# 9. Reporting of Results

- Results will be reported as:
  - $\circ$  Mean  $\pm$  SD
  - o Mean difference (95% CI)
  - o p-values and effect sizes
- Graphical presentations may include:
  - o ISI pre-post boxplots
  - o Sleep onset latency distributions
  - Sleep efficiency comparison plots
  - Sleep hypnogram examples

# 10. Deviations from the Statistical Analysis Plan

Any deviations from this SAP will be:

- Documented with justification
- Approved prior to final database lock
- Clearly described in final reports and publications

P.6